CLINICAL TRIAL: NCT05754567
Title: CONCEPTT Kids International Neurodevelopmental Outcomes Among Offspring of Women With Type 1 Diabetes: A Follow up Study of the CONCEPTT Randomized Control Trial
Brief Title: CONCEPTT Kids International Neurodevelopmental Outcomes Among Offspring of Women With Type 1 Diabetes
Acronym: CONCEPTTKids
Status: Recruiting | Type: Observational
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); SRI International (Industry)
Responsible Party: Sponsor
Other Study IDs: 4178
Record Dates: First submitted 2023-02-13; First posted 2023-03-06 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-12

CONDITIONS: Neurocognitive Disorders
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Neurodevelopmental Outcomes among Offspring of women with Type 1 Diabetes: A Follow up Study of the CONCEPTT Randomized Control Trial (CONCEPTT Kids International). An international, multicentre prospective cohort study of child and mother pairs. The potential number of recruits is 225 and the main inclusion criteria is child's mother who participated in the CONCEPTT Trial.

DETAILED DESCRIPTION:
This is a multicentre, international prospective cohort study of child and mother pairs from sites in Canada, UK, Spain and Italy. The expected duration of the study is three years. Women who participated in CONCEPTT will be invited to participate in CONCEPTT Kids International. Once informed consent is obtained, mothers will be asked to complete forms and questionnaires that provide information on family socio-demographics and their children's executive functions and behaviour (i.e. social responsiveness and attention). Self-reported height and weight measures of the child and parent(s) will also be collected.

Our primary outcome measure is childhood executive function measured by the Global Executive Composite of the Behaviour Rating Inventory of Executive Function - Second Edition (BRIEF2)

The secondary outcome measures were chosen based on our systematic review and meta-analysis, which identified significant associations between maternal pre-existing diabetes, and ASD and ADHD. We will use two parent-completed questionnaires to assess symptoms associated with these disorders; the Social Responsiveness Scale-2 (SRS-2) for behaviours associated with ASD and the ADHD Rating Scale-5 (ADHD-5) for ADHD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Children of women who participated in the CONCEPTT trial at selected recruiting sites

Exclusion Criteria:

* NA

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Children, ages 6 and up, of women with T1D who participated in the CONCEPTT trial
Sampling Method: Non-Probability Sample
Enrollment: 225 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Childhood executive function | 15 minutes
  The BRIEF2 (Behaviour Rating Inventory of Executive Function - Second Edition) is a parent-report 63 item questionnaire will be utilized to measure of executive function in school-aged children and adolescents (5-18 years of age). The BRIEF2 (Behaviour Rating Inventory of Executive Function - Second Edition) provides three broad index scores (i.e., Behaviour Regulation, Emotional Regulation, and Cognitive Regulation) and a General Executive Composite score. Results are provided in the form of T scores (mean=50, SD=10) with higher scores indicative of greater executive function difficulties; T scores of 65 are considered clinically elevated and indicative of executive function deficits.

SECONDARY OUTCOMES:
Significant associations between maternal pre-existing diabetes and ASD (Autism Spectrum Disorder) | 15 minutes
  The secondary outcome measures were chosen based on our systematic review and meta-analysis, which identified significant associations between maternal pre-existing diabetes and ASD (Autism Spectrum Disorder). The investigators will use a parent-completed questionnaire; the Social Responsiveness Scale-2 (SRS-2) for behaviours associated with ASD (Autism Spectrum Disorder).
Significant associations between maternal pre-existing diabetes and ADHD (Attention Deficit Hyperactivity Disorder) | 15 minutes
  The secondary outcome measures were chosen based on our systematic review and meta-analysis, which identified significant associations between maternal pre-existing diabetes and ADHD (Attention Deficit Hyperactivity Disorder). The investigators will use a parent-completed questionnaire; the ADHD Rating Scale-5 (ADHD-5) for ADHD (Attention Deficit Hyperactivity Disorder) symptoms.

OTHER OUTCOMES:
Maternal CGM (Continuous Glucose Monitor) percentage time in target | through study completion, an average of 2 year
  Primary Exposure: Maternal CGM (Continuous Glucose Monitor) percentage time in target range (3.5-7.8 mmol/L) during pregnancy. CGM (Continuous Glucose Monitor) percentage time in target range was chosen because it is the most accurate measure of fetal exposure to maternal glycemia during pregnancy. Additionally, percentage time in range has been associated with important neonatal outcomes such as neonatal hypoglycemia.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Alberta Health Services, Calgary, Alberta
  - IWK Health, Halifax, Nova Scotia
  - Mt Sinai Hospital, Toronto, Ontario